CLINICAL TRIAL: NCT01642316
Title: The Effect of Washback on Reading Comprehension
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nazila zarghi, faculty member, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: reading comprehension
Record Dates: First submitted 2012-07-11; First posted 2012-07-17 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2008-10

CONDITIONS: Reading Comprehension
Keywords: washback, reading comprehension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- washback (Experimental): students received 8 specific related formative test for that lesson plus a pre-test and post-test, Michigan English language proficiency test
  Interventions: Other: washback
- control (Other): students only received two tests, Michigan test of English language proficiency as pre-test and post-test.
  Interventions: Other: routin intervention

INTERVENTIONS:
Other: washback — students received 8 specific related formative test for that lesson. plus a pre-test and post-test, Michigan English language proficiency test
  Arms: washback
Other: routin intervention — students only received two tests, Michigan test of English language proficiency as pre-test and post-test.
  Arms: control

SUMMARY:
Testing and teaching are completely interrelated in education process; using various kinds of tests teachers are able to anticipate about the strong and weak points of learning in students, their progress and their accomplishment. The influence a test on teaching and learning is commonly referred to as washback. Testing washback is a twisted concept that becomes even more complex under a various interpretations of the washback phenomenon on teaching and learning. This study aimed to describe washback behaviors of students, in the low stakes testing in an ESP environment in two-fold. First, the study investigated the effects of different formative tests on Iranian medical students' English reading comprehension achievement. Secondly, the study explores the effects of washback on the students' attitudes toward English reading comprehension. The pre- and post-tests and one questionnaire were used to collect the data from Iranian medical students. Data were analyzed by paired t-test, t-test, and Mann-Whitney U test.

ELIGIBILITY:
Inclusion Criteria:

* nursing students
* study at mums

Exclusion Criteria:

* other disciplines
* study at other universities

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
improving reading comprehension | up to one year
  improving reading comprehension scored by Michigan Test of English Proficiency